CLINICAL TRIAL: NCT06288022
Title: Comparison of Total Tubeless Mini-PCNL Versus Tubeless Mini-PCNL : A Randomized Controlled Trial
Brief Title: Comparison of Total Tubeless Mini-PCNL Versus Tubeless Mini-PCNL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Thanakorn Sirajarus, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COA. MURA2023/947
Record Dates: First submitted 2024-02-24; First posted 2024-03-01 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Surgery-Complications; Nephrolithiasis Staghorn Calculus; Safety Issues
Keywords: total tubeless PCNL; complication; safety; tubeless PCNL
MeSH Terms: conditions — Staghorn Calculi

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial in 2 group
  1. total tubeless mini-PCNL
  2. tubeless mini-PCNL
Who Masked: Participant, Care Provider
Masking Description: All eligible patients will be provided with an explanation of the research and invited to participate.
  Patient will participate or not depends on whether they not meet the surgical exclusion criteria. If they meet the criteria, they will not participate in the research. If they not meet the criteria, they will be randomly assigned to one of the groups.
  Patients will not be informed of the treatment intervention in advance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- total tubeless mini-PCNL (Experimental): When finish the mini-PCNL operation, patient not receive placement both ureteral drainage tube (DJ-stent) and nephrostomy tube.
  Interventions: Other: total tubeless mini-PCNL
- tubeless mini-PCNL (Active Comparator): When finish the mini-PCNL operation, patient receive placement ureteral drainage tube (DJ-stent) but not receive nephrostomy tube.
  Interventions: Other: tubeless mini-PCNL

INTERVENTIONS:
Other: total tubeless mini-PCNL — When finish the mini-PCNL operation, patient not receive placement both ureteral drainage tube (DJ-stent) and nephrostomy tube.
  Arms: total tubeless mini-PCNL
Other: tubeless mini-PCNL — When finish the mini-PCNL operation, patient receive placement ureteral drainage tube (DJ-stent) but not receive nephrostomy tube.
  Arms: tubeless mini-PCNL

SUMMARY:
Limited literature has focused on the use of totally tubeless mini-percutaneous nephrolithotomy (Mini-PCNL) for the treatment of large renal stones.

This Randomized Controlled trial aims to compare complication and safety of Mini-PCNL between total tubeless and tubeless Mini-PCNL.

DETAILED DESCRIPTION:
After being informed about study and potential risks, all patient giving written informed consent with undergo a mini-PCNL operation. Patient who meet the eligibility requirements will be randomized in a single-blind manner (patient) in a 1:1 ratio to total tubeless mini-PCNL or tubeless mini-PCNL.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with kidney stones with a size ranging from 20 to 40 millimeters.
* Patients have undergone mini-PCNL, unilateral
* Absence of urinary tract infections before surgery.
* No urological congenital abnormality
* No coagulopathy

Exclusion Criteria:

* Presence of residual stones after the surgery, fragments larger than 4 millimeters.
* Patients with a single functioning kidney
* Complicated cases, including:

  1. massive bleeding in the upper tract during surgery
  2. Severe collecting systems injury during surgery
  3. Severe UPJ mucosa swelling considered unsafe by the physician, requiring the placement of a DJ stent or nephostomy tube
* Participants who decline or request withdrawal from the research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
incidence of complications between total tubeless mini-pcnl and tubeless mini-PCNL | from post operative day 0 to day 45
  The main objective is to study the incidence of complications between total tubeless mini-pcnl and tubeless mini-PCNL

SECONDARY OUTCOMES:
The secondary objective is to assess the surgical outcomes between total tubeless mini-pcnl and tubeless mini-PCNL | from post operative day 0 to day 45
  surgical outcomes such as bleeding, post operative pain, length of hospital stay, stone free rate.

CONTACTS AND LOCATIONS:
Overall Officials: THANAKORN SIRAJARUS, Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Ramathibodi Hospital, Mahidol University, Bangkok, Ratchathewi, Thailand

IPD SHARING:
Plan to Share IPD: No